CLINICAL TRIAL: NCT04294420
Title: Patient Education in Children and Adolescents With Pain-predominant Functional Gastrointestinal Disorders: a Pilot Study
Brief Title: Patient Education in Children With Functional Gastrointestinal Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Agneta Uusijärvi, Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-05417
Record Dates: First submitted 2020-02-25; First posted 2020-03-04 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient education program (Experimental): Patient education program
  Interventions: Behavioral: Patient education program

INTERVENTIONS:
Behavioral: Patient education program — The education program provides information and guidance concerning aetiology, diagnostics and treatment of pain-predominant functional gastrointestinal disorders. The patient education program will be provided in a group setting and the children will participate along with one of their parents. The participants (n=20) will be divided into two groups consisting of ten child-parent pairs. Two lectures will be held, two weeks apart, two hours per lecture. Represented teachers are physician, psychologist and dietician.

SUMMARY:
This pilot-study aims to evaluate the effect size and feasibility of patient education for children and adolescents (age 8-17 years) with pain-predominant functional gastrointestinal disorders (irritable bowel syndrome, functional abdominal pain and functional dyspepsia according to the Rome III criteria).

DETAILED DESCRIPTION:
The patient education will be provided in a group setting and the children will participate along with one of their parents. Education consists of 2-hour long group sessions, given at 2 different occasions within a month.

The hypothesis is that patient education will reduce gastrointestinal symptoms and pain and also improve quality of life in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents between 8-17 years (until their 18th birthday) who have been diagnosed with any of the diagnoses irritable bowel syndrome, functional dyspepsia or functional abdominal pain according to the Rome III criteria.
* Blood samples, with normal outcome, in terms of complete blood count (CBC), Erythrocyte Sedimentation Rate (ESR), Anti-tissue Transglutaminase Antibody (tTG), and dipstick urinalysis. Faecal Calprotectin should be measured if diarrhea is present.

Exclusion Criteria:

* Insufficient skills in the Swedish language.
* Severe psychiatric comorbidity (as suicidality, psychosis etc).
* Severe somatic comorbidity.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Treatment acceptability | Baseline to 3 months.
  A questionnaire to child /adolescent if they found the education logic. If they believe it will decrease symptoms. If they would recommend it to others

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory Gastrointestinal Symptoms Scales (PedsQL Gastro) | Baseline to 3 months, baseline to 6 months.
  Change in gastrointestinal symptoms measured with with a 14-item scale ranging from 0 (never) to 4 (almost always) measured from baseline to three months and from baseline to six months for analysis of effect. Improvements yield increased values.
Rome IV Diagnostic Questionnaire on Pediatric Functional Gastrointestinal Disorders (R4PDQ) | Baseline to 3 months, baseline to 6 months.
  Change in children's functional gastrointestinal disorders diagnostic status measured by Rome IV Diagnostic Questionnaire on Pediatric Functional Gastrointestinal Disorders (R4PDQ) - Child: Non-numerical self-report form for Children and Adolescents (10 years and older) measured from baseline to three months and from baseline to six months for analysis of effect as a self-rating scale from baseline to three months and from baseline to six months for analysis of effect.
Faces Pain Rating Scale. (FACES) | Baseline to 3 months, baseline to 6 months.
  Change in pain intensity measured with a self-rating scale daily during two weeks at baseline, daily during two weeks after 3 months and daily during two weeks after 6 months for analysis of effect. The Faces Pain Scale is a self-report measure used to assess the intensity of children's pain. Faces have four faces representing least pain and most pain on equal intervals on a scale from 0 (no pain)-10 (worst pain). Its validity is supported by a strong positive correlation (r=0.93, N=76) with a visual analogue scale (VAS) measure in children aged 5-12 years. The metric for scoring (0-10) conforms closely to a linear interval scale.Higher scores indicates higher levels of pain.
Pediatric Quality of Life Inventory (PedsQL) | Baseline to 3 months, baseline to 6 months.
  Change in quality of life from baseline to three months and from baseline to six months measured with a self-report scale that measures quality of life in adolescents. PedsQL Generic Core scales is a 23-item scale ranging from 0 (never) to 4 (almost always). Improvements yield increased values. The PedsQL is shown to distinguish between healthy children and adolescents and pediatric patients with acute or chronic health conditions and demonstrate acceptable reliability and validity.
The behavioral responses questionnaire child-adapted short scale (BRQ-C) | Baseline to 3 months, baseline to 6 months.
  Change in Gastrointestinal symptom-specific behaviors measured with a self-rating scale from baseline to three months and from baseline to 6 months, for analysis of effect. The BRQ-C comprise 11 items on a 7 point-scale, with only endpoints defined: never (0) and always (7). Higher scores indicates higher levels of gastrointestinal symptoms.
Children's Somatization Inventory (CSI-24) - subscale for gastrointestinal symptoms (CSI gastro) | Baseline to 3 months, baseline to 6 months.
  A questionnaire that assesses the perceived severity of 24 nonspecific somatic symptoms. Items are based off of the symptom criteria for somatization disorders as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM). We will use the subscale for gastrointestinal symptoms (CSI gastro) with questions concerning presence of gastrointestinal symptoms measured with a 7-item scale ranging from 0 (not at all) to 4 (very much) measured from baseline to three months and from baseline to six months. Higher scores indicates higher levels of somatization.
Spence Children Anxiety Scale - short version (SCAS-S) | Baseline to 3 months, baseline to 6 months.
  The SCAS-S assesses anxiety in children. The frequency of anxiety symptoms is rated on a 4-point scale, with answers ranging from never (0) to always (3). Higher scores indicates higher levels of anxiety. The SCAS-S will be assessed from baseline to three months and from baseline to six months.
Child Depression Inventory - short version (CDI-S) | Baseline to 3 months, baseline to 6 months.
  Child Depression Inventory (CDI) is a self-measure of child depression symptoms. The short version of the CDI (CDI-S) consists of 10 items graded from 0 (no symptoms) to 2 (severe symptoms). The questionnaire covers depressive symptoms such as self-blame, loss of appetite and insomnia. The CDI-S has shown high correlation to other measures of depression and should be considered a valid measure of depression symptoms. Symptoms measured from baseline to three months and from baseline to six months. Higher scores indicates higher levels of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Agneta Uusijärvi, MD PhD, Principal Investigator — Karolinska Institute, CLINTEC
Locations (1):
- Karolinka Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No